CLINICAL TRIAL: NCT05777564
Title: Tolerability of High Intensity Aerobic Exercise for Patients With Knee Osteoarthritis and Cardiovascular Disease Risk Factors
Brief Title: Tolerability of High Intensity Exercise for Knee Osteoarthritis
Acronym: THIPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Cecilie Bartholdy, Post Doc, Frederiksberg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-22064954
Record Dates: First submitted 2023-02-09; First posted 2023-03-21 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis; Cardiovascular Diseases
Keywords: knee osteoarthritis; cardiovasculare diseases; aerobic exercise; tolerance
MeSH Terms: conditions — Osteoarthritis, Knee; Cardiovascular Diseases | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: prospective study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT for knee OA (Other): high intensity exercise
  Interventions: Other: High intensity exercise

INTERVENTIONS:
Other: High intensity exercise — High intensity exercise on a indoor aerobic exercise device.

SUMMARY:
Background: Current knee osteoarthritis (OA) guidelines recommend knee specific exercise as treatment for knee OA pain. However, up to 87 % of patients with knee OA have at least one other chronic condition, typically cardiovascular in nature. The elevated risk of cardiovascular health problems can be mitigated by performing aerobic exercise. By consequence, it seems logical to apply aerobic exercise for this patient group as the symptomatic benefit is equal to other types of exercise.

Aim: This study aims to assess the tolerability of cardiovascular exercise using High Intensity Interval Training (HIIT) on different self-selected exercise equipment in patients with knee OA and at least one CVD risk factor.

Hypothesis: The hypothesis is that performing HIIT exercise is tolerable when having knee OA and at least one CVD risk factor.

Method:

The study is a prospective cohort study designed to assess if HIIT performed by patients with knee OA and at least one modifiable CVD risk factor influence knee pain. The investigators plan to include 40 participants. The participants will be recruited from the osteoarthritis outpatient clinic at Bispebjerg-Frederiksberg hospital.

This study will include participants with a clinical diagnosis of knee OA (either one or both knees) and at least one CVD risk factor (obesity, hypertension, elevated HbA1c (long-term blood glycose), elevated triglycerides, elevated cholesterol (LDL)). All participants will attend the HIIT intervention 3 times per week, for 12 weeks. Before a participant attend their first exercise session, he/she will be asked to complete an educational session about knee OA and aerobic exercise.

Participants will have a pre-screening visit (phone call), a screening visit, and a baseline visit, before the 12-week exercise period (3 sessions weekly), and after completion of the exercise period a follow-up visit.

Finance: This study is fully funded by Sygesikring "Denmark".

Publication: All results, both negative, positive, and inconclusive will be published. Should publication fail, the results will be made publicly available.

DETAILED DESCRIPTION:
BACKGROUND Current knee osteoarthritis (OA) treatment guidelines recommend knee specific exercise as treatment for knee OA pain. If performed regularly, such knee-specific exercise can yield a small to moderate effect on knee OA pain. However, muscle strengthening and neuromuscular exercise are not the only types of exercise that can reduce knee pain; walking regularly or aerobic exercise have similar positive effects on knee OA pain.

Up to 87 % of patients with knee OA have at least one other chronic condition. In the OA population abdominal obesity and metabolic syndrome are more prevalent than in the general population and knee OA is associated with increased risk for all-cause and cardiovascular (CV) death.

It therefore seems logical to apply aerobic exercise for this patient group as the symptomatic benefit is equal to other types of exercise.

AIM This study aims to assess the tolerability of cardiovascular exercise using High Intensity Interval Training (HIIT) on different self-selected exercise equipment in patients with knee OA and at least one CVD risk factor.

STUDY DESIGN The study is a prospective cohort study designed to assess if High Intensity Interval Training (HIIT) performed by patients with knee OA and at least one modifiable CVD risk factor influence knee pain.

The intervention will be performed with 3 sessions per week for 12 weeks. Due to the feasibility-like nature of this study, we have not made formalized sample size calculations. Approaches to the sample size justification for feasibility studies vary greatly. We plan to include 40 participants, whom we believe are adequate to meet the aims of the study and inform recruitment and sample size estimation for a subsequent large-scale randomized controlled trial. The participants will be recruited from the osteoarthritis outpatient clinic at Bispebjerg-Frederiksberg hospital. Participants that have completed the baseline visit will not be replaced if they are prematurely terminated or withdraw study participation.

DIAGNOSIS This study will include participants with a clinical diagnosis of knee OA (either one or both knees) and at least one CVD risk factor (obesity, hypertension, elevated HbA1c (long-term blood glycose), elevated triglycerides, elevated cholesterol (LDL)).

STUDY TREATMENT, HIIT All participants will attend the HIIT intervention 3 times per week, for 12 weeks and one educational session. The educational session containing information on rationale for aerobic exercise in knee OA and management of potential knee OA symptom flares. The educational session will be led by health professionals with experience within the fields of aerobic exercise and knee OA.

There will be several types of exercise equipment for aerobic exercise available (e.g., treadmill, cross-trainer, etc.) and participants will be asked to choose which they preferrer. If, during the intervention period, participants change exercise equipment (either due to pain or personal preference) this will be noted. There is no limit to the number of modalities a participant may chose.

Resistance (speed, watt, and/or elevation) will be regulated continuously throughout the intervention period to ensure the protocolized perceived exertion level are met at each exercise session.

TREATMENT ADHERENCE Attendance to each session will be recorded as participants meeting at the gym. Completion of the exercise sessions will be registered as perceived exertion (Borg) during the intervals, total time on the exercise equipment, hearth rate monitoring, speed, and resistance.

CONCOMITANT THERAPY All concomitant medications and treatments for knee OA should be kept stable during study participation and will be recorded in the study database. During the exercise period participants will be asked if the change their use of pain medication (increase/decrease dose) and this will be registered.

PARTICIPANT SAFETY The study personnel and clinical staff will monitor each participant for evidence of adverse event (AEs) throughout the study. The study personnel will assess and record any AE in detail including the date of onset, description, severity, duration and outcome, relation of the AE to study treatment, and any action(s) taken. In addition, a work-EKG will be measured at the baseline-visit to ensure the HIIT-protocol is safe for the participant (se Cardiopulmonary exercise test (VO¬2peak)).

Discontinuation of the entire study

The research group that initiated this study has the right to terminate this study at any time. Reasons may include the following, but are not restricted to:

• The incidence of events in this or other studies that indicate a potential health hazard to participants.

STUDY VISITS All consenting participants will undergo screening (assessment of eligibility), fill out questionnaires, have a clinical examination, a blood sample drawn, and perform a cardiovascular fitness test (VO¬2peak) before starting the exercise program. These initial assessments will be repeated at the last study visit. All participants will attend the clinic once for an educational session, and 3-weekly exercise sessions for 12 weeks.

Study completion The end-of-study is defined as the date of the last participant's last scheduled visit or the actual date of follow-up contact, whichever is the longer.

DETERMINATION OF SAMPLESIZE AND STATISTICAL ANALYSIS PLAN Determination of sample size This study is designed to assess tolerance of the purposed aerobic exercise intervention and therefore, no sample size is performed. A convenience sample of 40 participant is considered adequate to assess the tolerance of the study intervention and inform recruitment and sample size estimation for a subsequent large-scale randomized controlled trial.

Statistical consideration The statistical analyses will be described in detail in a statistical analysis plan to be completed before the last participant's last visit. For assessment of the aim (tolerance) all participants included in the study (completion of baseline visit) will be counted in the summation of results (intention-to-treat principle). If relevant, scores will be presented as mean/median with lower and upper limits. Occurrence of AEs will be reported in detail. The statistical tests of change for KOOS, VO¬2peak, blood sample outcomes, weight, and blood pressure will be two-sided and statistical significance will be claimed if the computed p-value is equal to or lower than 0.05.

RESEARCH ETHICS All participants are informed of their rights to withdraw from the study at any time without this impacting on any future investigations and/or treatments at any site or by some of the members of the study group.

After information is delivered, read, and understood, voluntary informed consent is given by the participants by signing a consent form before study participation can take placePrior to consent, it must be ensured that a potential participant have been given sufficient time to consider his or her participation.

Aerobic exercise at high intensities can cause discomfort due to breathlessness, which is why trained health professional are present at each exercise session to help guide participants through the sessions and observe if any unexpected reactions occur. Breathlessness is necessary for the exercise intervention to have an effect on the cardiopulmonary system. Symptomatic flares (knee pain) are not unlikely to occur during the first period of the exercise program, but these are expected to subside as the participant and his/her knee get accustomed to the exercise program. The participants will be fully informed about this aspect of the intervention. If participants are uncomfortable or experience unexpected reactions to the exercises the health professional present will react professionally and provide best care for the participant and refer to medical examination if judged necessary.

Health research ethical approval This protocol, the informed consent form, written patient information, any anticipate advertising materials, and relevant supporting information will be submitted to the health research ethical committee system by the study coordinator (Cecilie Bartholdy) prior to study initiation. The study will be conducted in accordance with the Danish law, the Helsinki declaration, and health research ethics committee requirements. The study coordinator is responsible for keeping the committee informed of amendments or changes to the protocol, and the progress of the study, as appropriate.

SOURCE DOCUMENTS AND DATABASES This research study group/institution will permit study-related monitoring, audits, and regulatory inspection(s) access to source data documents.

Study database This study will use an in-house custom-built electronic study database and an in-house custom-built electronic data capture system (Cirkeline). The applications meet all regulatory standards and allow management of all activities related to a clinical study, ensuring optimal resource use and safety according to good clinical practice and data protection legislation.

REGULATORY STANDARDS Participant confidentiality Participants medical information obtained by this study is confidential, and disclosure to third parties other than those noted below is prohibited.

If data from this study are published, the presentation format will not include names, recognizable photos, personal information, or other data which compromises the anonymity of participating participants.

Data Protection Act and General Data Protection Regulation The study will be conducted in accordance with the Data Protection Act and follow the General Data Protection Regulation. The study data management and data security procedures will be approved by the Regional Knowledge Center on Data Protection Compliance (videnscenter for dataanmeldelser i Region Hovedstaden).

Quality assurance All data will be entered into a study database for analysis and reporting. Any data captured electronically will be stored electronically in a separate database according to standard procedures at the Parker Institute. Upon completion of data entry, the database will be checked to ensure acceptable accuracy and completeness. System backups and record retention for the study data will be consistent with the Parker Institute standard procedures.

Financing and insurance information The study is initiated by Professor Marius Henriksen and post doc Cecilie Bartholdy who have received full funding from Sygeforsikringen "danmark" for the specific purpose to complete this study and a subsequent randomized controlled trial (total 5.6 mio DKK). None from the research group have conflicts of interests related to the funding of this study. This information is disclosed to all participants in the written information material.

All sources of support (including technical and financial) provided for this study is disclosed in the written information material and in publication of the study results. All future financial and/or technical support to the study is disclosed to alle participants (previous, current, and potential) in the written information material.

The participants are insured by the Danish Patient Insurance Association. Financing and insurance issues are addressed in the written information material.

PUBLICATION Development of the core publication will be coordinated by the research group, that consist of people who have provided significant input into study design, implementation, conduct, and interpretation as recommended by the international committee of medical journal editors (ICMJE).

I accordance with the principles of the Helsinki Declaration, all results in this study, positive as well as negative, and inconclusive will be published. If publication, for any given reason fails, the results will be made publicly available.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with knee OA
* At least one of the following CVD risk factors: Overweight/obesity, hypertension, elevated HbA1c, elevated triglycerides, High LDL
* Age > 18
* Willing and able to understand and participate in the study

Exclusion Criteria:

* Contraindication to exercise (e.g. resting systolic blood pressure > 200 or diastolic blood pressure > 115, acute or reoccurring chest pain)
* Major cardiovascular event within the last 5 years
* Planning to start another treatment for their knee OA during the study participation period
* Performing at least 150 minutes of moderate intensity activities or ≥ 75 minutes of vigorous activity weekly
* Insulin dependent type I or type II diabetes
* Scheduled surgery during study participation
* Evidence of other inflammatory joint disease (e.g., rheumatoid arthritis or gout)
* Generalized pain syndromes such as fibromyalgia
* Lumbar or cervical nerve root compression syndromes
* Other musculoskeletal, neurological, or medical condition precluding participation to aerobic exercise
* Any other condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or which obstruct participation, such as a large knee joint effusion, uncontrolled diabetes/hypertension, psychiatric disorders, or opiate dependency.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Knee flares | from exercise week 1-12
  number of knee flares reported during the exercise period, a flare is defined at an increase of minimum 2 on a numeric rating scale from 0-10
Average knee pain | from exercise week 1-12
  reported average knee pain from first to last exercise session on a numeric rating scale from 0-10
Attendance | from exercise week 1-12
  number of attended sessions during the exercise period

SECONDARY OUTCOMES:
Completion of the HIIT protocol | from exercise week 1-12
  number of exercise sessions where the HIIT protocol is completed as described will be recorded
Cardiopulmonary test (Vo2peak) | at baseline (week 0) and after completion of the exercise period (week 13)
  Measurement of peak oxygen consumption
Knee Injury and Osteoarthritis Outcome Score (KOOS) | baseline (week 0) and follow-up (week 13)
  measure of knee related quality of life, using the subgroups: pain, symptoms, activities of daily living, sport and recreation, knee related quality of life.
PainDETECT Questionnaire | baseline (week 0)
  tool for the assessment of the patient pain. The questionnaire consist of seven sensory symptoms items, one temporal item, and one spatial item. Finally, three measure of knee pain: current knee pain, past 4-week strongest knee pain and average past 4-week knee pain
Blood sample (cholesterol) | baseline (week 0) and follow-up (week 13)
  A fasting blood sample will be collected to measure cholesterol (LDL).
Blood sample (triglycerides) | baseline (week 0) and follow-up (week 13)
  A fasting blood sample will be collected to measure triglycerides
Blood sample, HbA1c | baseline (week 0) and follow-up (week 13)
  A fasting blood sample will be collected to measure HbA1c
Blood pressure | baseline (week 0) and follow-up (week 13)
  Systolic and diastolic blood pressures are measured using a standard blood pressure apparatus
Weight | baseline (week 0) and follow-up (week 13)
  weight will be measured on a digital weight.
Analgesics use | baseline (week 0) and follow-up (week 13)
  Participant reported use of paracetamol and ibuprofen at baseline and last study visit recorded by the study personnel

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Bartholdy, PhD, Principal Investigator — The Parker Institute, Frederiksberg Hospital
Locations (1):
- The Parker Insitute, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request from another research party all data can be made avaliable.
Supporting Information: Study Protocol, SAP
Time Frame: The SAP will become available at clincialtrials.gov before last patient last visit. The study protocol will be available if requested. Upon reasonable request from other researchers, addition data will be made available.
Access Criteria: The request must be from an established research group. Approved ethical and data management documents must obtained before data sharing is accommodated.